CLINICAL TRIAL: NCT06292793
Title: Cyclical Sighing for Pain in an Orthopedic Clinic Waiting Room
Brief Title: Cyclical Sighing for Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00004696
Record Dates: First submitted 2023-12-13; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Coping Information (Active Comparator)
  Interventions: Behavioral: Pain Coping Information
- Cyclical Sighing (Experimental)
  Interventions: Behavioral: Cyclical Sighing

INTERVENTIONS:
Behavioral: Pain Coping Information — A 4-minute audio recording providing common pain coping techniques (e.g., ice, rest, medication, surgery).
  Arms: Pain Coping Information
Behavioral: Cyclical Sighing — A 4-minute audio recording consisting of a 1-minute introduction to cyclical sighing followed by a 3-minute cyclical sighing practice.
  Arms: Cyclical Sighing

SUMMARY:
This is a single-site, two-arm, parallel-group randomized clinical trial (RCT). The clinical effects of a 4-minute audio-recorded cyclical sighing intervention for orthopedic patients will be investigated relative to a 4-minute audio-recoding about pain psychoeducation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Seeking treatment at the Tallahassee Orthopedic Clinic

Exclusion Criteria:

* Cognitive impairment preventing completion of study procedures.
* Other unstable illness judged by medical staff to interfere with study involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | immediately after the 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most unpleasant pain imaginable.

SECONDARY OUTCOMES:
Change in Pain Intensity Numeric Rating Scale | Immediately after the 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most intense pain imaginable.
Change in Anxiety Numeric Rating Scale | Immediately after the 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no anxiety and 10 representing intense anxiety.
Change in Depression Numeric Rating Scale | Immediately after the 4-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no depression and 10 representing intense depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Tallahassee Orthopedic Clinic (TOC), Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hanley AW, Davis A, Worts P, Pratscher S. Cyclic sighing in the clinic waiting room may decrease pain: results from a pilot randomized controlled trial. J Behav Med. 2025 Apr;48(2):385-393. doi: 10.1007/s10865-024-00548-5. Epub 2025 Feb 4. PMID 39904867